CLINICAL TRIAL: NCT00092456
Title: Comparison of the Immunogenicity and Safety of Three Consistency Lots of V260 in Healthy Infants
Brief Title: Consistency Lots Vaccine Study (V260-009)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-009; 2004_078
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Rotavirus Infections
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines; RotaTeq

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- RotaTeq™ Lot 1 (Experimental): ~8.81 X 10^7 IU/Dose of RotaTeq™
  Interventions: Biological: rotavirus vaccine, live, oral, pentavalent
- RotaTeq™ Lot 2 (Experimental): ~8.01 X 10^7 IU/Dose of RotaTeq™
  Interventions: Biological: rotavirus vaccine, live, oral, pentavalent
- RotaTeq™ Lot 3 (Experimental): ~6.91 X 10^7 IU/Dose of RotaTeq™
  Interventions: Biological: rotavirus vaccine, live, oral, pentavalent
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rotavirus vaccine, live, oral, pentavalent — Three oral doses (~8.81 X 10^7 IU/Dose for Lot 1; ~8.01 X 10^7 IU/Dose for Lot 2; and ~6.91 X 10^7 IU/Dose for Lot 3) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination
  Other Names: V260; RotaTeq™
  Arms: RotaTeq™ Lot 1; RotaTeq™ Lot 2; RotaTeq™ Lot 3
Biological: Placebo — Placebo-matching RotaTeq™ administered at 3 separate visits scheduled 4 to 10
  weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination
  Arms: Placebo

SUMMARY:
This study was designed to evaluate consistency in the antibody response to three manufactured lots of an investigational Rotavirus Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants

Exclusion Criteria:

* History of abdominal disorders from a birth defect, intussusception, or abdominal surgery
* Known or suspected problems with the immune system
* Fever at time of immunization
* Prior administration of a rotavirus vaccine
* History of known prior rotavirus disease, chronic diarrhea, or failure to thrive.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 793 (Actual)
Dates: Start 2003-05; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 sites in the United States from 09-May-2003 (first patient in) to 02-Jul-2004
  (last dose given).
  Last subject completed follow-up: 13-Aug-2004.
  All data corrections applied (Frozen File) date: 30-Sep-2004
Pre-assignment Details: Subjects with prior rotavirus disease, chronic diarrhea, and fever at time of immunization were excluded
  from the trial.
Groups:
- RotaTeq™ Lot 1: Three oral doses (~8.81 X 10^7 IU/Dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination.
- RotaTeq™ Lot 2: Three oral doses (~8.01 X 10^7 IU/Dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination.
- RotaTeq™ Lot 3: Three oral doses (~6.91 X 10^7 IU/Dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination.
Period: Overall Study
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Started | 226 (Subject assigned to ~8.81 X 10^7 IU/Dose of RotaTeq™ - Lot 1) | 225 (Subject assigned to ~8.01 X 10^7 IU/Dose of RotaTeq™ - Lot 2) | 229 (Subject assigned to ~6.91 X 10^7 IU/Dose of RotaTeq™ - Lot 3) | 113 (Subjects assigned to Placebo-matching RotaTeq™)
Vaccinated at Visit 1 | 226 | 225 | 229 | 113
Vaccinated at Visit 2 | 208 | 217 | 210 | 104
Vaccinated at Visit 3 | 202 | 210 | 200 | 98
Completed | 201 (Subjects who received 3 scheduled vaccinations; with up to 42 days safety follow-up after each dose) | 208 (Subjects who received 3 scheduled vaccinations; with up to 42 days safety follow-up after each dose) | 200 (Subjects who received 3 scheduled vaccinations; with up to 42 days safety follow-up after each dose) | 97 (Subjects who received 3 scheduled vaccinations; with up to 42 days safety follow-up after each dose)
Not Completed | 25 | 17 | 29 | 16
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — Protocol Violation | 5 | 7 | 8 | 6
Not completed — Withdrawal by Subject | 13 | 5 | 16 | 6
Not completed — Moved | 1 | 1 | 0 | 1
Not completed — Other | 4 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- RotaTeq™ Lot 2: Three oral doses ( ~8.01 X 10^7 IU/Dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination.
- RotaTeq™ Lot 3: Three oral doses ( ~6.91 X 10^7 IU/Dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow up after each vaccination.
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo | Total
Number analyzed (Participants) | 226 | 225 | 229 | 113 | 793
Age, Customized [Number; unit: participants]
  6 to 12 Weeks | 225 | 224 | 228 | 113 | 790
  Over 12 Weeks | 1 | 1 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 98 | 108 | 43 | 367
  Male | 108 | 127 | 121 | 70 | 426
Race/Ethnicity, Customized [Number; unit: participants]
  White | 139 | 144 | 147 | 68 | 498
  Hispanic American | 57 | 49 | 52 | 28 | 186
  Black | 13 | 11 | 6 | 5 | 35
  Multi-Racial | 10 | 10 | 16 | 6 | 42
  Other | 7 | 11 | 8 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Serum Neutralizing Antibodies (SNA) Response Against Rotavirus Serotypes G1, G2, G3, G4 and P1A[8]
Description: Antibody response to 3 manufactured lots of RotaTeq™ and placebo groups, based on the SNA PostDose 3 geometric mean titers (GMTs) (expressed in dilution units) against rotavirus serotypes G1, G2, G3, G4 and P1A[8]
Time Frame: 42 days following the 3rd vaccination
Population: Per Protocol Population; excluding protocol violators and subjects with invalid data based on laboratory determinations.
Measure: Geometric Mean (95% Confidence Interval); unit: dilution units
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 225 | 229 | 113
dilution units
  G1 SNA (dilution units) | 167.9 [135.7 to 207.7] | 193.2 [157.6 to 236.8] | 171.0 [140.6 to 208.1] | 9.3 [7.2 to 11.9]
  G2 SNA (dilution units) | 20.7 [17.3 to 24.7] | 22.6 [19.1 to 26.8] | 17.8 [15.1 to 20.9] | 5.9 [5.3 to 6.6]
  G3 SNA (dilution units) | 18.0 [15.2 to 21.2] | 18.5 [15.7 to 21.9] | 14.6 [12.4 to 17.2] | 9.6 [7.4 to 12.5]
  G4 SNA (dilution units) | 66.0 [57.0 to 76.4] | 74.3 [64.4 to 85.7] | 65.7 [55.6 to 77.5] | 7.8 [6.5 to 9.4]
  P1A[8] SNA (dilution units) | 71.1 [60.0 to 84.2] | 72.3 [61.4 to 85.3] | 65.6 [55.0 to 78.2] | 10.2 [7.6 to 13.5]
Statistical Analysis 1: Comparison: RotaTeq™ Lot 1 vs RotaTeq™ Lot 2; A pairwise comparison of lots was made for each serotype, for each pair of lots; Test type: Non-Inferiority or Equivalence — If equivalence was established in all 3 pairwise comparisons for a given serotype, the 3 lots were considered consistent for that serotype. Each comparison consisted of 2 one-sided tests of equivalence with α=0.05. Statistical significance for the 2 one-sided equivalence tests for each pair of lots was established if the p-values for the hypothesis tests were each less than 0.05. This corresponds to the 2-sided 90% CI for the fold difference in the 2 lots being contained entirely within (0.5,2); p < 0.001, ANOVA — The reported p-value is for all 5 serotypes, no multiplicity adjustment made, and Type I error rate controlled at the 0.05 level. P<0.05 implies that the difference is statistically significantly less than the prespecified difference of 2 fold
Statistical Analysis 2: Comparison: RotaTeq™ Lot 1 vs RotaTeq™ Lot 3; A pairwise comparison of lots was made for each serotype, for each pair of lots; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: RotaTeq™ Lot 2 vs RotaTeq™ Lot 3; A pairwise comparison of lots was made for each serotype, for each pair of lots; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Other Pre Specified Outcome: Geometric Mean Antibody Titer(s) (GMT) to Serum Anti-rotavirus Immunoglobulin A (IgA).
Description: Post Dose 3 serum samples were assayed for serum anti-rotavirus IgA
Time Frame: 42 days following the 3rd vaccination
Population: Per Protocol Population; excluding protocol violators and subjects with invalid data based on laboratory determinations.
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 225 | 229 | 113
units/mL | 292.7 [241.0 to 355.5] | 272.5 [227.9 to 325.7] | 266.2 [220.1 to 321.8] | 0.4 [0.2 to 0.8]

3. Other Pre Specified Outcome: Number of Subjects With Clinical Adverse Experiences (CAEs)
Description: Subjects in this study were followed for all CAEs, including intussusception. A CAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: Up to 42 days following each study vaccination, or until the time of the subsequent study vaccination(s), whichever occurred first
Population: Safety Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  With CAEs | 207 | 213 | 212 | 101
  Without CAEs | 19 | 11 | 17 | 10

4. Other Pre Specified Outcome: Number of Subjects With Serious Clinical Adverse Experiences (SCAEs)
Description: Subjects were followed for all SCAEs. SCAEs are any CAEs occurring at any dose that: results in death; or is life threatening; or results in persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is cancer; or is an overdose.
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  With Serious CAEs | 4 | 4 | 2 | 3
  Without Serious CAEs | 222 | 220 | 227 | 108

5. Other Pre Specified Outcome: Number of Subjects With Vaccine-Related Clinical AEs (CAEs)
Description: CAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product. Vaccine-related CAEs are CAEs that are assessed by an investigator, who is a qualified physician, as being related to the vaccine according to his/her best clinical judgment.
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  With vaccine-related CAEs | 167 | 173 | 165 | 78
  Without vaccine-related CAEs | 59 | 51 | 64 | 33

6. Other Pre Specified Outcome: Number of Subjects With Serious Vaccine-Related Clinical AEs (CAEs)
Description: Serious vaccine-related CAEs are CAEs assessed by an investigator as being related to the vaccine that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is cancer; or is an overdose
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  With serious vaccine-related CAEs | 0 | 0 | 0 | 1
  Without serious vaccine-related CAEs | 226 | 224 | 229 | 110

7. Other Pre Specified Outcome: Number of Subjects Discontinued Due to Clinical Adverse Experiences
Description: A CAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  Discontinued due to CAEs | 0 | 0 | 1 | 1
  Not discontinued due to CAEs | 226 | 224 | 228 | 110

8. Other Pre Specified Outcome: Number of Subjects Discontinued Due to Vaccine-Related Clinical Adverse Experiences (CAEs)
Description: CAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product. Vaccine-related CAEs are CAEs that are assessed by an investigator who is a qualified physician as being related to the vaccine according to his/her best clinical judgment.
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  Discontinued due to vaccine-related CAEs | 0 | 0 | 0 | 1
  Not discontinued due to vaccine-related CAEs | 226 | 224 | 229 | 110

9. Other Pre Specified Outcome: Number of Subjects Discontinued Due to Serious Clinical Adverse Experiences (SCAEs)
Description: SCAEs are any CAEs that: results in death; or is life threatening; or results in persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is cancer; or is an overdose.
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  Discontinued due to serious CAEs | 0 | 0 | 1 | 1
  Not discontinued due to serious CAEs | 226 | 224 | 228 | 110

10. Other Pre Specified Outcome: Number of Subjects Discontinued Due to Serious Vaccine-related Clinical Adverse Experiences (CAEs)
Description: as for outcome 6
Time Frame: as for outcome 3
Population: All subjects who were vaccinated and followed up
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Number analyzed (Participants) | 226 | 224 | 229 | 111
Participants
  Discontinued due to serious vaccine-related CAEs | 0 | 0 | 0 | 1
  NOTdiscontinued dueto serious vaccine-related CAEs | 226 | 224 | 229 | 110

ADVERSE EVENTS:
Time Frame: Patients in this study were followed for all adverse experiences, for up to 42 days following each study vaccination, or until the time of the subsequent study vaccination(s), whichever occurred first.
Description: The number of patients listed in the Adverse Event tables (226 - Lot 1, 224 - Lot 2, 229 - Lot 3, and 112 - Placebo) is the number of patients who received study treatment.
  Although a patient may have had two or more clinical adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | RotaTeq™ Lot 1 | RotaTeq™ Lot 2 | RotaTeq™ Lot 3 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/226 | 4/224 | 2/229 | 3/111
Other Adverse Events (participants affected / at risk) | 206/226 | 212/224 | 211/229 | 101/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ Lot 1 (N=226) | RotaTeq™ Lot 2 (N=224) | RotaTeq™ Lot 3 (N=229) | Placebo (N=111)
Congenital ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 2 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ Lot 1 (N=226) | RotaTeq™ Lot 2 (N=224) | RotaTeq™ Lot 3 (N=229) | Placebo (N=111)
Ear pain (Ear and labyrinth disorders) | 2 | 4 | 0 | 0
Conjunctivitis (Eye disorders) | 14 | 10 | 9 | 7
Dacryostenosis acquired (Eye disorders) | 2 | 2 | 8 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 8 | 15 | 7
Diarrhoea (Gastrointestinal disorders) | 110 | 122 | 103 | 50
Flatulence (Gastrointestinal disorders) | 10 | 16 | 11 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 6 | 8 | 1
Infantile colic (Gastrointestinal disorders) | 5 | 5 | 2 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Regurgitation of food (Gastrointestinal disorders) | 5 | 3 | 2 | 0
Teething (Gastrointestinal disorders) | 1 | 4 | 5 | 0
Vomiting (Gastrointestinal disorders) | 74 | 85 | 77 | 34
Injection site discomfort (General disorders) | 6 | 8 | 6 | 6
Injection site pain (General disorders) | 14 | 27 | 20 | 7
Pyrexia (General disorders) | 119 | 122 | 115 | 52
Hypersensitivity (Immune system disorders) | 1 | 3 | 2 | 0
Bronchiolitis (Infections and infestations) | 16 | 14 | 21 | 7
Bronchitis (Infections and infestations) | 4 | 2 | 3 | 0
Candida nappy rash (Infections and infestations) | 5 | 2 | 1 | 3
Croup infectious (Infections and infestations) | 3 | 6 | 4 | 2
Ear infection (Infections and infestations) | 2 | 6 | 4 | 2
Eye infection (Infections and infestations) | 1 | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 11 | 7 | 7 | 3
Herpangina (Infections and infestations) | 1 | 1 | 3 | 0
Impetigo (Infections and infestations) | 0 | 1 | 2 | 2
Influenza (Infections and infestations) | 2 | 5 | 3 | 3
Nasopharyngitis (Infections and infestations) | 40 | 50 | 34 | 22
Oral candidiasis (Infections and infestations) | 10 | 8 | 7 | 6
Otitis media (Infections and infestations) | 46 | 53 | 51 | 20
Pharyngitis (Infections and infestations) | 1 | 1 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 3 | 2 | 0
Rhinitis (Infections and infestations) | 4 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 73 | 71 | 69 | 36
Viral infection (Infections and infestations) | 4 | 13 | 6 | 4
Viral rash (Infections and infestations) | 3 | 2 | 4 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 5 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 3 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9 | 12 | 3
Agitation (Psychiatric disorders) | 4 | 3 | 1 | 2
Crying (Psychiatric disorders) | 3 | 1 | 4 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 3 | 0
Irritability (Psychiatric disorders) | 31 | 49 | 49 | 18
Sleep disorder (Psychiatric disorders) | 1 | 3 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 23 | 29 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 27 | 20 | 22 | 11
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 9 | 11 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 4 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 6 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 6 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 8 | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.